CLINICAL TRIAL: NCT04713449
Title: Enhancing Self Care Among Oral Cancer Survivors: The Empowered Survivor Trial
Brief Title: Enhancing Self Care Among Oral Cancer Survivors: The Empowered Survival Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Cancer Registry of Greater California (Unknown); The New Jersey State Cancer Registry (Unknown)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Chief, Behavioral Sciences, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 132004; Pro2020000768 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Oral Cancer; Oropharyngeal Cancer; Head and Neck Cancer
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowered Survivor online (Experimental): The online intervention, called Empowered Survivor (ES) is a self-management intervention for patients with head and neck cancer. The intervention contains the following modules: Introduction; Difficulty Swallowing and Muscle Strength; Oral Care; Long-term Follow-Up Care/Oral exams; Calm and Connect; and Maintaining.
  Interventions: Other: Empowered Survivor Online; Other: Survey Administration
- Springboard Beyond Cancer (Active Comparator): Springboard Beyond Cancer is a general resource for survivors of all cancer. It is a free self-management program for cancer survivors developed by trusted sources, the ACS and the NCI.
  Interventions: Other: Springboard Beyond Cancer; Other: Survey Administration

INTERVENTIONS:
Other: Empowered Survivor Online — Informational online intervention for head and neck cancer survivors
  Arms: Empowered Survivor online
Other: Springboard Beyond Cancer — Informational online intervention for all cancer survivors
  Arms: Springboard Beyond Cancer
Other: Survey Administration — Survey measures administered at BL, two and 6 months post-baseline

SUMMARY:
Project's goal is evaluate an online tool the research team created called Empowered Survivor (ES) against a free online self-management intervention developed for cancer survivors by the National Cancer Institute and the American Cancer Society called Springboard Beyond Cancer.

DETAILED DESCRIPTION:
600 patients who have completed treatment between one and three years ago and are currently cancer-free will be recruited via the New Jersey State Cancer Registry or the Cancer Registry of Greater California and randomly assigned to ES or Springboard Beyond Cancer. Participants will complete measures at baseline, 2, and 6-months post-baseline. The investigators will also complete a process evaluation of Empowered Survivor.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* Diagnosed with a first primary invasive oral or oropharyngeal cancer between 1 and 3 years ago;
* Currently cancer free (but can have experienced a recurrence);
* Has internet access;
* Read English;
* Has sufficient vision to read a survey and complete an online intervention

Exclusion Criteria:

-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Self-efficacy score | Baseline, two and 6 months post-baseline
  Change in self- efficacy measured with the Self-efficacy scale (22 items) which targets confidence in managing aspects of self-care (e.g., dry mouth, swallowing, oral self-exam, communicating with providers, emotions). Administered at multiple time points to measure effect of the intervention. Ratings range from 1 (not at all confident) to 5 (very confident). An item average will be calculated.
Preparedness for survivorship | Baseline, two and 6 months post-baseline
  Change in preparedness for survivorship. The Preparedness for survivorship scale (10 items) developed by the investigator assesses whether information received about survivorship was sufficient, helpful, comprehensive, and covered self-care tasks. Administered at multiple time points to measure effect of the intervention. Items are rated on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree). Higher score indicate better preparedness.
Quality of Life score measured using the The European Organization for Research and Treatment of Cancer (EORTC)- Head and Neck | Baseline, two and 6 months post-baseline
  Change in QOL score over time. The European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire- Head and Neck-43. The European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire- Head and Neck-43 is the updated version of the EORTC H&N 35, used in the researcher's pilot work. The EORTC QLQ-HN is the most widely-used measure of Head and Neck QOL. The investigators use the total score in analyses, but will evaluate subscales. Administered at multiple time points to measure effect of the intervention. Items are rated on 1 (not at all)-4 (very much) Likert scale and higher scores indicate worse QOL.

SECONDARY OUTCOMES:
Performance of oral self-exam, past month | Baseline, two and 6 months post-baseline
  1 item asking the participant if he/she has performed an oral self-exam, past month. Yes/No. Administered at multiple time points to measure effect of the intervention.
Comprehensiveness is the number of areas checked (11 areas) during the oral self-exam | Baseline, two and 6 months post-baseline
  Change in comprehensiveness of exams over time. 11 items will list the areas to check and ask participant to indicate Yes/No if the participant checked that area during the oral self-exam. Administered at multiple time points to measure effect of the intervention.
Performance of exercises to improve swallowing, past month (yes/no) | Baseline, two and 6 months post-baseline
  One question asking participants if they have completed exercises to improve swallowing in the past month. Administered at multiple time points to measure effect of the intervention.
Performance of head/neck exercises, past month (yes/no) | Baseline, two and 6 months post-baseline
  One question asking participants if they have completed head and neck exercises in the past month. Administered at multiple time points to measure effect of the intervention.

OTHER OUTCOMES:
Action and Planning Coping | Baseline, two and 6 months post-baseline
  Change in Action and Planning coping score. The scale (8 items) assesses the degree to which a detailed plan is made for self-care tasks. Administered at multiple time points to measure effect of the intervention. Items are rated on a 5-point Likert scale(1 = strongly disagree, 5 = strongly agree). Mean scale score will be reported. Higher score = higher action coping.
Patient activation | Baseline, two and 6 months post-baseline
  Change in Patient activation scale score. Patient Activation Scale (13 items) assesses the active role in cancer care. Administered at multiple time points to measure effect of the intervention. Items are rated on a 4-point scale (1 = Disagree strongly, 4 = Agree strongly). Higher score = higher activation.
Information Needs | Baseline, two and 6 months post-baseline
  Change in score over time. Information needs (23 items) is adapted from the FOCUS Health-Related Topics measure. Administered at multiple time points to measure effect of the intervention. Participants reported if they would like more information on each topic (yes/no). The number of " yes" responses are averaged.
Support needs | Baseline, two and 6 months post-baseline
  Change in Support needs. The support needs scale (34 items) assesses physical, psychological, and health care needs. Administered at multiple time points to measure effect of the intervention. Participants are asked to indicate the extent to which they needed help in the past month (1 = No Need; Not applicable, "This is not a problem",2 = No need; Satisfied, "I did need help but my need was satisfied," 3 = Low need; "It caused me concern and I had little need for additional help," 4 = Moderate need-"It caused me concern and I had some need for additional help," 5 = High need; -"It caused me concern and I had a strong need for additional help"). Support needs that are rated as "moderate"(4) or "high" need (5) will be summed, with a range of 0 to 34.
Concerns about recurrence scale | Baseline, two and 6 months post-baseline
  Change in concerns about recurrence. The first 4 items from the concerns about recurrence scale are measured on a 1-6 scale. with lower scores indicating less concerns or worry. The additional 21 items are rated on 0 (not at all) to 4 (extremely) with higher scores indicating more concerns or worry. Administered at multiple time points to measure effect of the intervention.
Moderator-Race/ethnicity | Baseline only
  Race/ethnicity will be assessed.
Moderator-Receipt of survivorship care plan | Baseline only
  Yes/No did the participant receive a survivorship care plan
Moderator- Baseline self-efficacy score | Baseline Only
  The baseline score on the scale will be (22 items) examined. The scale targets confidence in managing aspects of self-care (e.g., dry mouth, swallowing, oral self-exam, communicating with providers, emotions). Ratings are 1- 5

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manne SL, Imanguli M, Kashy D, Pesanelli M, Frederick S, Van Cleave JH, Paddock L, Hudson S, Steinberg M, Clifford P, Domider M, Singh N. Enhancing Self-care Among Oral Cancer Survivors: Protocol for the Empowered Survivor Trial. JMIR Res Protoc. 2023 Jan 20;12:e39996. doi: 10.2196/39996. PMID 36662561

DOCUMENTS (1):
  • Informed Consent Form (2024-05-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT04713449/ICF_000.pdf